CLINICAL TRIAL: NCT03987555
Title: Pilot Feasibility Study of Paclitaxel Therapeutic Drug Monitoring in Cancer Patients
Brief Title: Paclitaxel Therapeutic Drug Monitoring in Cancer Patients
Status: Recruiting | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00058758; WFBCCC 01319 (Other: Wake Forest Baptist Comprehensive Cancer Center); P30CA012197 (NIH); NCI-2019-05616 (Other: National Cancer Institute)
Record Dates: First submitted 2019-06-13; First posted 2019-06-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumor, Adult; Metastatic Nonsmall Cell Lung Cancer; Anatomic Stage IV Breast Cancer AJCC v8; Metastatic Cervical Carcinoma; Metastatic Ovarian Carcinoma; Malignant Uterine Neoplasm; Vulvar Cancer; Invasive Breast Cancer; Metastatic Breast Carcinoma; Prognostic Stage IV Breast Cancer AJCC v8; Recurrent Breast Carcinoma; Recurrent Cervical Carcinoma; Recurrent Lung Non-Small Cell Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Vulvar Carcinoma; Stage IV Cervical Cancer AJCC v8; Stage IV Lung Cancer AJCC v8; Stage IV Vulvar Cancer AJCC v8; Stage IV Ovarian Cancer AJCC v8; Stage IVA Cervical Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVA Ovarian Cancer AJCC v8; Stage IVA Vulvar Cancer AJCC v8; Stage IVB Cervical Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8; Stage IVB Ovarian Cancer AJCC v8; Stage IVB Vulvar Cancer AJCC v8; Vulva Squamous Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Uterine Cervical Neoplasms; Ovarian Neoplasms; Uterine Neoplasms; Vulvar Neoplasms; Breast Neoplasms; Lung Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood draw for peripheral blood mononuclear cell isolation and subsequent use in pharmacogenomic assays.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood draws — Blood draws for serum and peripheral blood mononuclear cell isolation collected throughout treatment course
Other: QLQ-CIPN20 Survey — 20-item self-reported survey for participant reported symptoms related to chemotherapy-induced peripheral neuropathy
Other: PR-CTCAE Survey — 124-item survey addressing chemotherapy-induced peripheral neuropathy concerning severity of the numbness and tingling and the degree these symptoms interfere with daily activities.

SUMMARY:
The goals of this prospective, observational cohort study are to determine the feasibility of implementing paclitaxel therapeutic drug monitoring for cancer patients and explore the relationship between paclitaxel drug exposure and the development of neuropathic symptoms.

This trial studies if paclitaxel can be consistently measured in the blood of patients with solid tumors undergoing paclitaxel treatment. Drugs used in chemotherapy, such as paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Nerve damage is one of the most common and severe side effects of paclitaxel. The ability to consistently measure paclitaxel in the blood may allow doctors to control the dose of paclitaxel, so that enough chemotherapy is given to kill the cancer, but the side effect of nerve damage is reduced.

DETAILED DESCRIPTION:
Primary Objective:

• Determine the feasibility of monitoring paclitaxel serum drug levels in patients with a solid tumor (e.g. lung, breast, and gynecologic cancers) for which Paclitaxel is the standard of care.

Secondary Objectives:

* Compare Paclitaxel serum drug levels among patients with differing degrees of chemotherapy-induced peripheral neuropathy at the end of Paclitaxel treatment.
* Compare mitochondrial function within circulating peripheral blood mononuclear cells among patients with differing degrees of chemotherapy-induced peripheral neuropathy at the end of Paclitaxel treatment.
* Compare the ability of pulsed electromagnetic field to modulate immune cells of individuals experiencing differing degrees of chemotherapy-induced peripheral neuropathy at the end of Paclitaxel treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female sex
* Age ≥ 18 years
* Individuals receiving treatment at the Wake Forest Comprehensive Cancer Center who are anticipated to receive paclitaxel for curative or palliative intent, with or without surgery and/or radiation (i.e. neoadjuvant, adjuvant, or in the setting of recurrent or metastatic disease) as per decision with their medical oncologist for the following malignancies and dosing regimens:
* Invasive breast cancer (any HER2 and ER/PR status)
* Patients considered for curative or palliative chemotherapy with paclitaxel 80-175 mg/m2 with or without doxorubicin, cyclophosphamide, carboplatin, trastuzumab, bevacizumab, or pertuzumab

Cervical cancer • Patients considered for curative or palliative chemotherapy with paclitaxel 135-175 mg/m2 with or without cisplatin, carboplatin, topotecan, or bevacizumab

Non-small cell lung cancer

• Patients considered for curative or palliative chemotherapy with paclitaxel 45-200 mg/m2 with or without carboplatin, cisplatin, bevacizumab, atezolizumab, or pembrolizumab

Ovarian cancer • Patients considered for curative or palliative chemotherapy with paclitaxel 60-175 mg/m2 with or without carboplatin, cisplatin, ifosfamide, gemcitabine, pazopanib, or bevacizumab

Uterine neoplasms

• Patients considered for curative or palliative chemotherapy with paclitaxel 135-175 mg/m2 with or without carboplatin, cisplatin, doxorubicin, ifosfamide, bevacizumab, or trastuzumab

Vulvar cancer (squamous cell carcinoma)

* Patients considered for curative or palliative chemotherapy with paclitaxel 60-175 mg/m2 with or without cisplatin, carboplatin, or bevacizumab
* Ability to understand and the willingness to sign an IRB-approved informed consent document (either directly or via a legally authorized representative)
* Patients with prior radiation treatment or surgery will not be disqualified from enrollment into the study, unless the aforementioned interventions resulted in peripheral neuropathy as a complication

Exclusion Criteria:

* Prior treatment with PTX, for any duration or indication
* Prior treatment with neurotoxic chemotherapy including any taxane, vinca alkaloid, platinum-containing agent, bortezomib, or thalidomide that has resulted in clinical symptoms of persistent, CTCAE grade II or higher peripheral neuropathy
* Concurrent enrollment in a clinical study of a neuroprotective intervention at the time of study initiation
* Any contraindication to Paclitaxel (e.g. history of allergic reaction to paclitaxel or Kolliphor EL)
* Current signs or symptoms of peripheral neuropathy at the time of enrollment, e.g. due to diabetes, HIV, or other conditions
* Known personal or family history of hereditary peripheral neuropathy (e.g. Charcot-Marie-Tooth disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is designed to enroll male and female patients with histologically-confirmed solid tumors who are anticipated to receive Paclitaxel as part of the curative or palliative antineoplastic therapy. The study will target lung, breast, and gynecologic (i.e. cervical, ovarian, uterine, and vulvar) cancers specifically.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-11-11 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants Completing Paclitaxel Infusions | One day after last infusion dose
  Feasibility will be assessed based on the proportion of patients who complete study blood draws at >90% of completed Paclitaxel infusions. A completed Paclitaxel infusion is defined as each dose of Paclitaxel that is completed in its entirety. The a priori success rate will be defined as 90% of patients receiving 100% of study blood draws and the null rate will be set at 50%

SECONDARY OUTCOMES:
Differences in Maximum Plasma Concentration of Paclitaxel from Baseline to Completion | 30 days after completion of chemotherapy treatment
  Differences in descriptive characteristics (e.g. mean, median, standard deviation, etc.) of the Paclitaxel maximum plasma concentration (Cmax) among patients with and without chemotherapy-induced peripheral neuropathy according to the physician reported neuropathy CTCAE (Grade II or greater) at baseline and at the end of Paclitaxel treatment.
Differences in Time Above Threshold from Baseline to Completion | 30 days after completion of chemotherapy treatment
  Differences in descriptive characteristics (e.g. mean, median, standard deviation, etc.) of time above threshold (Tc>0.05) among patients with and without chemotherapy-induced peripheral neuropathy according to the physician reported neuropathy CTCAE (Grade II or greater) at baseline and at the end of Paclitaxel treatment.
Differences in Inflammasome Activation from Baseline to Completion | 30 days after completion of chemotherapy treatment
  Differences in inflammasome activation following pulsed electromagnetic field stimulation between patients with and without chemotherapy-induced peripheral neuropathy according to the physician reported neuropathy CTCAE at baseline and at the end of Paclitaxel treatment.
Differences in Inflammatory Cytokine Production from Baseline to Completion | 30 days after completion of chemotherapy treatment
  Differences in inflammatory cytokine production following pulsed electromagnetic field stimulation between patients with and without chemotherapy-induced peripheral neuropathy according to the physician reported neuropathy CTCAE at baseline and at the end of Paclitaxel treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Roy Strowd, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No